CLINICAL TRIAL: NCT05936060
Title: Recovery of Joint Cartilage in Adults With Knee Osteoarthritis by Use of Mesenchymal Stromal Cells Derived From Human Umbilical Cord: Randomized Controlled Clinal Trial With Clinical and Radiologic Outcomes
Brief Title: Cartilage Recovery in Adults With Knee Osteorthritis by Mesenchymal Cell Therapy: Randomized Trial of Radiologic and Clinical Outcomes
Acronym: INMUNOCEM-OA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GUSTAVO SALGUERO (Other)
Collaborators: Hospital Infantil Universitario de San Jose (Other)
Responsible Party: Sponsor-Investigator, GUSTAVO SALGUERO, Research Leader Advanced Therapies Unit, Instituto Distrital de Ciencia, Biotecnología e Innovación en Salud - IDCBIS
Organization: Instituto Distrital de Ciencia, Biotecnología e Innovación en Salud - IDCBIS (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDCBIS-UTA-EC-01-InmunoCEM
Record Dates: First submitted 2023-06-16; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMUNOCEM (Experimental): Administration of umbilical cord-derived mesenchymal stromal cells suspension
  Interventions: Biological: INMUNOCEM
- PLASMALYTE (Placebo Comparator): Administration of plasmalyte as vehicle for MSC
  Interventions: Drug: PLACEBO COMPARATOR

INTERVENTIONS:
Biological: INMUNOCEM — Mesenchymal Stromal Cell suspension intraarticularly injected
  Other Names: Mesenchymal stromal cell suspension
  Arms: IMUNOCEM
Drug: PLACEBO COMPARATOR — Administration of plasmalyte as a vehicle for MSC
  Other Names: PLASMALYTE
  Arms: PLASMALYTE

SUMMARY:
The treatment of osteoarthritis (OA) of the knee remains still controversial. Despite that fact advanced stages with symptomatic and functional improvement are obtained with total knee replacement, however, there is no treatment that neither modifies the natural history of this disease, nor avoid joint replacement surgery in young patients in whom the prosthesis has conflictive indications. Moreover, prosthetic surgery leads to lower long-term survival and in older patients, higher morbidity and mortality. Cell therapy promises to be a treatment option through the use of mesenchymal cells with the capacity control inflammatory responses and trigger the differentiation into chondrocytes. Here we propose a randomized placebo-controlled clinical trial to evaluate radiologic and clinical outcomes in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

Pain most days for the last month. Presence of osteophytes. Synovial fluid with mechanical characteristics. Morning stiffness for less than 30 minutes in the affected joint. Patellar crepitus. Patients aged 40 years or older and less than 60 years. Radiological criteria for osteoarthritis of the knee Kellgren-Lawrence 2 to 4 in comparative radiographs with knee support taken in the last 12 months prior to consultation.

Pain in one or both knees according to a visual analogue scale of 5 or more, out of 10 points in the last 3 months.

Exclusion Criteria:

Consumption of non-steroidal anti-inflammatory drugs or anticoagulants in the last 14 days.

Patient with a history of joint infiltration or arthroscopic surgery of the affected knee in the last 6 months.

Participants in another treatment or research study within the past year. Pregnant or lactating patients. Patient with active tumor pathology or a history of oncological disease. Patient with metabolic disease and/or uncontrolled coagulopathy at the assessment time.

Patients who have received previous treatments such as microfractures, and osteochondral allografts.

Patients with present meniscal lesions. Patients with a history of thyroiditis or thyroid nodules with increased antithyroglobulin antibodies.

Patients with a history of osteoarticular infection in the last 5 years or active at the time of assessment.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Visual Analogue scale (VAS) | 30 months (day 0, day 1, month 1, month 3, month 6, year 1 and year 2
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between paints with similar conditions. Score ranges from 1 to 10, where 1 means lowest pain and 10 relates to highest pain
Changes in Knee Injury and Osteoarthritis Outcome Score (KOOS) | 30 months (day 0, month 3, month 6, year 1 and year 2)
  KOOS reflects the individual disease burden and overall joint health. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
Radiological changes in Magnetic resonance observation of cartilage repair tissue (MOCART 2.0) | 30 Months (day 0, year 1 and year 2)
  MOCART score was introduced based on 7 pertinent variables that facilitate a standardized, reproducible, semiquantitative approach for the morphological assessment of cartilage repair. Variables assesed in MOCART are: 1. Degree of cartilage defect; 2. integration into adjacent cartilage; 3. surface of the repair tissue; 4. structure of the repair tissue; 5. signal intensity of repaired tissue; 6. bony defect or bony overgrowth; 7. subchondral changes. The score ranges between 0 and 100, being 100 the maximum level of tissue compromise